CLINICAL TRIAL: NCT06914505
Title: Study on the Effectiveness and Safety of Visual Restoration Therapy in the Active Rehabilitation of Patients With Visual Field Defects
Brief Title: Study on the Effectiveness and Safety of VRT in Patients With Visual Field Defects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LYS2024211001
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Visual Field Defects; Visual Field Loss
Keywords: visual field defect; visual restoration therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VRT treatment group (Experimental): The participants will be provided with a pair of appropriate vision aids and will undergo 3 times 30-minute visual restoration therapy (VRT) training per week for three months.
  Interventions: Behavioral: visual restoration therapy
- control group (No Intervention): Participants will be provided with a pair of appropriate vision aids, however without any visual treatment.

INTERVENTIONS:
Behavioral: visual restoration therapy — In this study, we used a reversing checkerboard pattern as a stimulus and acted on the relatively dark spots area of the patient's visual field.
  Other Names: photostimulation therapy
  Arms: VRT treatment group

SUMMARY:
The goal of this clinical trial is to learn if visual restoration therapy (VRT) (a type of treatment that aims to improve vision) works to the visual rehabilitation of patients with visual field defects. It will also learn about the safety of VRT. The main questions it aims to answer are:

* Can visual reconstruction therapy help expand the visual field in patients with visual field defects?
* What medical problems do patients with visual field defects experience during the procedure of VRT? Researchers will look at how patients with visual field defects who use a visual aid in combination with VRT and those who use a visual aid only, compare the visual field expansion at three months to see how well visual reconstruction therapy works.

Participants will:

* will undergo a specialized visual function assessment and be provided with a pair of appropriate vision aids.
* Visit the clinic at one month and three months after enrolment for review of visual function and completion of a Chinese-version Low Vision Quality of Life (CLVQOL) questionnaire.
* Participants receiving VRT will additionally undergo 30 minutes of VRT three times per week for 3 months.
* Keep a diary for their symptoms and severity and frequency of occurrence during treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a clear diagnosis of visual field defects.
2. Participants were between 18 and 80 years of age (including borderline values);
3. Participants have been treated for their primary disease and conditions are stable;
4. Participants are not at significant risk of vision loss in the last three months;
5. Participants do not have planned intraocular surgery during the trial period；
6. Participants can understand the trial protocol and sign informed consent.

Exclusion Criteria:

1. Participants diagnosed as blindness;
2. Participants with a previous history of seizures or other psychiatric disorders;
3. Participants with cognitive impairments;
4. Participant's attention span is less than 30 minutes;
5. Participants had conditions such as significant ptosis or severe dry eye;
6. Participants who were in poor general health or who could not cooperate in completing the study protocol for some reasons such as transport.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
visual field mean deviation (MD) value | A total of 3 examinations were performed during the trial: before treatment, after 1 month of treatment, and after 3 months of treatment.
  using the Humphrey Field Analyzer 30-2 test to obtain MD values

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Li, MD. and PHD., Principal Investigator — Ophthalmology Department, Xuanwu Hospital，Capital Medical University

IPD SHARING:
Plan to Share IPD: No